CLINICAL TRIAL: NCT03616028
Title: The CONFORMAL Early Feasibility Study An Evaluation of the Safety and Performance of the Conformal Left Atrial Appendage Seal for Left Atrial Appendage Occlusion
Brief Title: The CONFORMAL Early Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Conformal Medical, Inc (Industry)
Collaborators: Yale Cardiovascular Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18-101
Record Dates: First submitted 2018-07-30; First posted 2018-08-06 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Non-valvular Atrial Fibrillation
MeSH Terms: interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, open-label, first-in-human study aimed at examining the performance of the CLAAS device for LAA closure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Non-valvular AF adults (Experimental): Left atrial appendage closure (LAAC) with the CLAAS device will be performed according to the device Instructions for Use, based on TEE, ICE and angiographic guidance, femoral venous access and inter-atrial septum crossing.
  Interventions: Device: left atrial appendage closure

INTERVENTIONS:
Device: left atrial appendage closure — Closure of the left atrial appendage (LAAC) is performed percutaneously. Implantation of the CLAAS device will be performed according to device specific instructions for use based on both TEE guidance, ICE and angiography, femoral access and inter-atrial septum crossing

SUMMARY:
An evaluation of the safety and performance of the Conformal Left Atrial Appendage Seal for Left Atrial Appendage Occlusion

DETAILED DESCRIPTION:
The Conformal Left Atrial Appendage Seal (CLAAS) Device is a permanent implant designed to occlude the left atrial appendage (LAA) to eliminate blood flow into and clot passage from the LAA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female aged ≥18 years
2. Documented non-valvular AF (paroxysmal, persistent, or permanent)
3. High risk of stroke or systemic embolism, defined as CHA2DS2-VASc score of ≥ 2 for men and ≥ 3 for women
4. The patient is recommended for oral anticoagulation therapy (OAC), but has an appropriate rationale to seek a non-pharmacologic alternative to chronic oral anticoagulation
5. The patient deemed appropriate for LAA closure by the Site P.I. and a non-interventional physician using an evidenced-based decision-making tool on oral anticoagulants consistent with standard of care.
6. The patient is willing and able to comply with the protocol-specified medication regimen and follow-up evaluations
7. The patient (or legally authorized representative, (where allowed)) has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

General Exclusion Criteria

1. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following the index procedure. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days prior to index procedure.
2. Anatomic conditions that would prevent performance of an LAA occlusion procedure (e.g., prior atrial septal defect [ASD] or patient foramen ovale [PFO] surgical repair or implanted closure device, or obliterated or ligated left atrial appendage)
3. Atrial fibrillation that is defined by a single occurrence or that is transient or reversible (e.g., secondary thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures)
4. Patients with a medical condition (other than atrial fibrillation) that mandates chronic oral anticoagulation (e.g., history of unprovoked deep vein thrombosis or pulmonary embolism, or mechanical heart valve)
5. History of bleeding diathesis or coagulopathy, or patients in whom antiplatelet and/or anticoagulant therapy is contraindicated
6. Active infection with bacteremia
7. Documented symptomatic carotid artery disease (>50% diameter stenosis with prior ipsilateral stroke or TIA) or known asymptomatic carotid artery disease (diameter stenosis of >70%)
8. Recent (within 30 days pre-procedure) or planned (within 60 days post-procedure) cardiac or non-cardiac interventional or surgical procedure
9. Recent (within 90 days pre-procedure) stroke or transient ischemic attack.
10. Recent (within 60 days pre-procedure) myocardial infarction
11. Vascular access precluding delivery of implant with catheter-based system
12. Severe heart failure (New York Heart Association Class III or IV)
13. Prior cardiac transplant, history of mitral valve replacement or transcatheter mitral valve intervention, or any mechanical valve implant
14. Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 (by the Modification of Diet in Renal Disease equation), or dialysis at the time of screening
15. Platelet count <75,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <3,000 cells/mm3
16. Patient has a known allergy, hypersensitivity or contraindication to aspirin, heparin, or device materials (e.g., nickel, titanium, gold) or that would preclude any P2Y12 inhibitor therapy, or the patient has contrast sensitivity that cannot be adequately pre-medicated
17. Current participation in another investigational drug or device study
18. Patient is a prisoner
19. Patient is unable to undergo general anesthesia
20. Known other medical illness or known history of substance abuse that may cause non-compliance with the protocol or protocol-specified medication regimen, confound the data interpretation, or is associated with a life expectancy of less than 2 years
21. Patient has a condition which precludes adequate transesophageal echocardiographic (TEE) assessment

Echocardiographic Exclusion Criteria

1. Left atrial appendage anatomy cannot accommodate the CLAAS device per manufacturer IFU
2. Intracardiac thrombus or dense spontaneous echo contrast, as visualized by TEE within 2 days prior to implant
3. Left ventricular ejection fraction (LVEF) <30%
4. Circumferential pericardial effusion >10 mm or symptomatic pericardial effusion, signs or symptoms of acute or chronic pericarditis, or evidence of tamponade physiology
5. Atrial septal defect that warrants closure
6. High risk patent foramen ovale (PFO), defined as an atrial septal aneurysm (exclusion >15 mm or length > 15 mm) or large shunt (early [within 3 beats] or substantial passage of bubbles)
7. Moderate or severe mitral valve stenosis (mitral valve area <1.5 cm2)
8. Complex atheroma with mobile plaque of the aorta
9. Patient has evidence of cardiac tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Freedom from major adverse events: | up to 45 days
  Major adverse events defined as: All cause mortality, ischemic stroke, systemic thromboembolism, device or procedure-related adverse events requiring open cardiac surgery or major endovascular intervention.

SECONDARY OUTCOMES:
Closure success | 45 days post procedure, 6 months, 12 months
  Device success followed by complete closure or peri-device residual leak ,/= 5mm in width on TEE (evaluated by independent core lab)
Major Adverse Events | 1year, 2 years, 3 years, 4 years, 5 years
  All cause mortality, ischemic stroke, systemic thromboembolism, device or procedure-related adverse events requiring open cardiac surgery or major endovascular intervention.

CONTACTS AND LOCATIONS:
Overall Officials: William A Gray, MD, Principal Investigator — Main Line Health Lankenae Heart Institute
Locations (11):
- United States (11):
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Pacific Heart Institute, Santa Monica, California
  - Catholic Medical Center, Manchester, New Hampshire
  - Mount Sinai, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Lankenau Heart Institute, Wynnewood, Pennsylvania
  - Erlanger Health System, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Institute, Austin, Texas
  - Baylor Scott & white Research Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No